CLINICAL TRIAL: NCT06022536
Title: SSS40 A Single-center, Randomized, Double-blind, Placebo-controlled Phase I Clinical Study of Single-dose, Dose-escalation Safety, Tolerability, Pharmacokinetics, and Immunogenicity in Healthy Chinese Subjects.
Brief Title: A Clinical Study of SSS40 in Healthy Chinese Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of Clinical Trials Center of Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSS-SSS40-UND-I-01
Record Dates: First submitted 2023-08-27; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single-dose , dose escalation, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1mg dose group (Experimental): The 1mg dose group is a low dose group and only safety and tolerability will be evaluated, pharmacokinetics and immunogenicity will not be evaluated, therefore one subject is planned to be enrolled.1mg SSS40 was injected subcutaneously on day1.
  Interventions: Drug: SSS40
- 3mg dose group (Experimental): Four subjects were included in the 3mg dose group (trial group: 3:1 placebo group).3mg SSS40/Placebo was injected subcutaneously on day1.
  Interventions: Drug: SSS40; Drug: Placebo
- 10mg、20mg、30mg、 45mg、60mg or 80mg dose group (Experimental): Sentinel dosing was used starting with the 10 mg group, with two subjects first enrolled and randomized 1:1 (test drug:placebo) for sentinel dosing, with sentinels participating in blinding, and then after the sentinel group had completed the 72-h safety assessment, the rest of the subjects in the group were randomized to receive dosing according to the test drug group versus the placebo group.10mg、20mg、30mg、 45mg、60mg or 80mg SSS40/Placebo was injected subcutaneously on day1.
  Interventions: Drug: SSS40; Drug: Placebo

INTERVENTIONS:
Drug: SSS40 — Subjects injected with SSS40
Drug: Placebo — Subjects injected with Placebo
  Arms: 10mg、20mg、30mg、 45mg、60mg or 80mg dose group; 3mg dose group

SUMMARY:
This is a single-center, randomized, double-blind, single-administration, escalating-dose, placebo-controlled, phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of SSS40 in healthy subjects in China.

A total of 8 subcutaneous dose groups were planned, including 1mg, 3mg, 10mg, 20mg, 30mg, 45mg, 60mg, 80mg. Starting from the 10mg group, a sentinel approach was adopted, whereby 2 subjects were first enrolled in the group, and randomized to the sentinel group in a 1:1 ratio (test drug:placebo), with the sentinels blinded, and then the remaining subjects in the group were randomized according to a 1:1 ratio (test drug:placebo), and the sentinel group was blinded. After completion of the 72-h safety assessment in the sentinel group, the remaining subjects in the group were randomized to receive the drug according to the test drug group and the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent form prior to the trial, volunteered to participate in the trial, and was willing and able to follow the study protocol for medications, tests, visits, and other related procedures;
* At the time of signing the informed consent form, the age of 18-45 years old (including both sides of the border), the proportion of female subjects is not less than 1/3 of the sample in the group;
* Men weighing not less than 50kg and women weighing not less than 45kg, with BMI within the range of 19.0~26.0 (both sides included) [BMI=Weight (kg)/Height (m2)]；
* Those who have no abnormalities or whose abnormalities are not clinically significant after assessment of vital signs, physical examination, routine blood, urine, blood biochemistry, coagulation, pregnancy test (women of childbearing age), 12-lead electrocardiogram (ECG), abdominal B-ultrasound, and thyroid function at the time of screening;
* Subjects and their spouses or partners do not plan to have children or donate sperm/eggs and are willing to use reliable contraception or are not of childbearing potential from the time of initiation of study drug use (14 days prior to study drug use for females) through 6 months post-dose. The female subject is not lactating and has a negative pregnancy test.

Exclusion Criteria:

* Prior history of allergies or sensitivities；
* Diseases or factors with abnormal clinical manifestations, including, but not limited to, neurological, cardiovascular, hematologic, hepatic cardiovascular, hematologic, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immune, skeletal system diseases or other factors. other factors；
* History of bone or joint disease, including but not limited to osteoarthritis, avascular necrosis, destructive joint disease, pathologic fractures, osteonecrosis, rheumatoid arthritis, lupus erythematosus or arthritis, pathologic fractures, osteonecrosis, rheumatoid arthritis, neuropathic arthritis, lupus erythematosus, or Inflammatory Joint Diseases；
* History of joint-related events, including but not limited to joint trauma, total joint replacement, meniscus or knee ligament injury (with or without surgical repair), joint infection, joint dislocation total joint replacement, meniscus or knee ligament injuries (with or without surgical repair), joint infections, joint dislocations etc.
* Those with a history of clinically significant peripheral neuropathy, sensory abnormalities, and dullness of sensation；
* Those with a history of autonomic neuropathy or diabetic neuropathy；
* Those who have undergone surgery within 3 months prior to screening or are scheduled for surgery during the trial period；
* Use of any prescription drugs, over-the-counter drugs, and supplements within 2 weeks prior to screening；
* Average daily smoking ≥5 cigarettes or equivalent in the 3 months prior to screening；
* Average weekly alcohol consumption in the 3 months prior to screening of more than 14 Alcohol Units (1 Alcohol Unit is equivalent to. 360 ml of beer or 45 ml of 40% alcohol by volume spirits or 150 ml of red wine) or a positive breath alcohol result Positive；
* Those vaccinated within 4 weeks prior to screening or scheduled to be vaccinated during the study or within 4 weeks of the end of the trial；
* Those who have participated in a clinical trial of any drug and used the test drug within 3 months prior to screening；
* Participated in blood donation or large blood loss (≥200 ml) within 3 months before screening；
* Those with known factors that significantly interfere with normal venous blood collection, such as a history of needle or blood fainting；
* Those with a positive urine drug screening test；
* Persons with a known history of substance abuse and/or drug intake.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2023-10-26 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 57 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Peak Plasma Concentration (Cmax) | up to 57 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | up to 57 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | up to 57 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

IPD SHARING:
Plan to Share IPD: No